CLINICAL TRIAL: NCT00268398
Title: Essai De Phase III De Chimiotherapie Par FOLFOX 4 Ou Par Une Succession FOLFOX 7 - FOLFIRI Chez Des Patients Ayant Des Metastases Resecables D'Origine Colorectale - MIROX
Brief Title: Combination Chemotherapy in Treating Patients With Colorectal Cancer and Resectable Metastases
Acronym: MIROX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000453815; GERCOR-C02-1; GERCOR-C02-1-MIROX; EU-20567; SANOFI-GERCOR-C02-1
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Colorectal Cancer; Metastatic Cancer; Chemotherapy
Keywords: adenocarcinoma of the colon; stage IV colon cancer; adenocarcinoma of the rectum; stage IV rectal cancer; resectable metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Irinotecan

ARMS (2):
- FOLFOX4 (Active Comparator)
  Interventions: Drug: oxaliplatin, folinic acid, fluorouracil
- FOLFOX7 followed by FOLFIRI (Experimental)
  Interventions: Drug: oxaliplatin, irinotecan, folinic acid, fluorouracil

INTERVENTIONS:
Drug: oxaliplatin, folinic acid, fluorouracil — folinic acid 200 mg/m² (day 1&2) oxaliplatin 85 mg/m² (day 1) bolus 5FU 400 mg/m² (day 1&2) continuous 5FU 600mg/m² (day 1 to 2)
  Arms: FOLFOX4
Drug: oxaliplatin, irinotecan, folinic acid, fluorouracil — FOLFOX7 folinic acid 400 mg/m² (day 1) oxaliplatin 130 mg/m² (day 1) continuous 5FU 3000mg/m² (day 1 to 2)
  FOLFIRI folinic acid 400 mg/m² (day 1) irinotecan 180 mg/m² (day 1) bolus 5FU 400 mg/m² (day 1) continuous 5FU 2400mg/m² (day 1 to 2)
  Arms: FOLFOX7 followed by FOLFIRI

SUMMARY:
PURPOSE: This randomized phase III trial is studying two different combination chemotherapy regimens to compare how well they work in treating patients with colorectal cancer and resectable metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the 2-year disease-free survival rate in patients treated with these regimens.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Compare the tolerability of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Compare the objective response rate, postoperative complication rate, and transfusing rate in patients having metastasis surgery,
* Determine the pharmacogenetics of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter phase III study. Patients are stratified according to prior chemotherapy (perioperative vs postoperative), prior treatment (surgery only vs radiotherapy with or without surgery), and Blumgart score (0-1 vs 2-3 vs 4-5). Patients are randomized to 1 of 2 treatment arms.

* Arm I (FOLFOX 4): Patients receive FOLFOX 4 combination chemotherapy comprising oxaliplatin 85mg/m² IV over 2 hours, leucovorin calcium IV over 2 hours, fluorouracil IV bolus /15min and fluorouracil continuously over 22 hours on day 1. Treatment repeats every 2 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (FOLFOX 7 and FOLFIRI): Patients receive FOLFOX 7 combination chemotherapy comprising high-dose oxaliplatin 130mg/m² IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours on days 1 and 2. Treatment repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive FOLFIRI combination chemotherapy comprising irinotecan hydrochloride 180mg/m² IV over 30-90 minutes and leucovorin calcium and fluorouracil IV bolus /15min on day 1, and fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients in both arms who have undergone prior resection of metastatic lesions may undergo surgery after 6 courses of chemotherapy or after chemotherapy is completed.

Quality of life is assessed at baseline and after courses 4, 8, and 12.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 284 patients will be accrued for this study.

ELIGIBILITY:
MAIN ELIGIBILITY CRITERIA

DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum
* Resectable or resected metastatic disease,

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Alkaline phosphatase ≤ 5 times upper limit of normal (ULN)
* Bilirubin ≤ 2 times normal
* Creatinine ≤ 135 mmol/L or creatinine clearance ≥ 60 mL/min
* SGOT and SGPT ≤ 3 times ULN
* No peripheral neuropathy that affects normal functions
* No unresolved complications from prior surgery

PRIOR CONCURRENT THERAPY:

* At least 1 year since prior FOLFOX 4 or FOLFIRI regimen in the adjuvant setting
* No concurrent participation in another clinical trial
* Recovered from prior therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2002-07; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 2-year

SECONDARY OUTCOMES:
Overall survival | 2-year, 3-year, 5-year
Tolerability | 2-year
Quality of life | 2-year
Pharmacogenetics | 2-year

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hebbar, MD, Study Chair — Centre Hospital Universitaire Hop Huriez
Locations (32):
- France (32):
  - Institut Sainte Catherine, Avignon
  - Hopital Duffaut, Avignon
  - C.H.G. Beauvais, Beauvais
  - Hopital Saint Andre, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier Docteur Duchenne, Boulogne-sur-Mer
  - Centre Hospitalier de Briey, Briey
  - Centre Regional Francois Baclesse, Caen
  - Hopital Louis Pasteur, Chartres
  - Hopital Beaujon, Clichy
  - Louis Mourier Hospital, Colombes
  - Clinique du Parc, Croix
  - Hopital Drevon, Dijon
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Hopital Saint - Louis, La Rochelle
  - Hopital Robert Boulin, Libourne
  - Polyclinique Du Bois, Lille
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Polyclinique des Quatre Pavillons, Lormont
  - Hopital Saint Joseph, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - Centre Hospitalier Intercommunal Le Raincy - Montfermeil, Montfermeil
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Saint Antoine, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Tenon, Paris
  - Hopital Haut Leveque, Pessac
  - Polyclinique De Courlancy, Reims
  - Clinique Specialise du Littoral-Cote d'Opale, Saint-Martin-Boulogne
  - Clinique Charcot, Sainte-Foy-lès-Lyon
  - C.H. Senlis, Senlis
  - Hopital Foch, Suresnes

REFERENCES:
- [Derived] Hamidou Z, Chibaudel B, Hebbar M, Hug de Larauze M, Andre T, Louvet C, Brusquant D, Garcia-Larnicol ML, de Gramont A, Bonnetain F. Time to Definitive Health-Related Quality of Life Score Deterioration in Patients with Resectable Metastatic Colorectal Cancer Treated with FOLFOX4 versus Sequential Dose-Dense FOLFOX7 followed by FOLFIRI: The MIROX Randomized Phase III Trial. PLoS One. 2016 Jun 16;11(6):e0157067. doi: 10.1371/journal.pone.0157067. eCollection 2016. PMID 27310205
- [Derived] Hebbar M, Chibaudel B, Andre T, Mineur L, Smith D, Louvet C, Dutel JL, Ychou M, Legoux JL, Mabro M, Faroux R, Auby D, Brusquant D, Khalil A, Truant S, Hadengue A, Dalban C, Gayet B, Paye F, Pruvot FR, Bonnetain F, Landi B, Flesch M, Carola E, Martin P, Vaillant E, de Gramont A; Group Cooperateur Multidisciplinaire en Oncologie (GERCOR) Group. FOLFOX4 versus sequential dose-dense FOLFOX7 followed by FOLFIRI in patients with resectable metastatic colorectal cancer (MIROX): a pragmatic approach to chemotherapy timing with perioperative or postoperative chemotherapy from an open-label, randomized phase III trial. Ann Oncol. 2015 Feb;26(2):340-7. doi: 10.1093/annonc/mdu539. Epub 2014 Nov 17. PMID 25403578